CLINICAL TRIAL: NCT01456039
Title: A Japanese Phase 1/2, Multicenter, Open-label Study to Assess the Efficacy, Tolerability, Safety and Pharmacokinetics of Romidepsin in Subjects With the Progressive or Relapsed Peripheral T-cell Lymphoma
Brief Title: A Japanese Phase 1/2 Study to Assess the Efficacy, Safety and Pharmacokinetics of Romidepsin in Patients With Peripheral T-cell Lymphoma (PTCL)
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Celgene (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ROMI-TCL-001
Record Dates: First submitted 2011-10-18; First posted 2011-10-20 (Estimated); Results first posted 2016-08-19 (Estimated); Last update posted 2019-02-11 (Actual); Status verified 2019-01

CONDITIONS: Lymphoma, T-cell, Peripheral
MeSH Terms: conditions — Lymphoma, T-Cell, Peripheral | interventions — romidepsin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Romidepsin (Experimental): Patients will receive romidepsin intravenously for 4 hours on Days 1, 8, and 15 of each 28-day cycle until when/if a discontinuation criterion, e.g., disease progression, severe adverse events, or consent withdrawal.
  Interventions: Drug: Romidepsin

INTERVENTIONS:
Drug: Romidepsin — Intravenous dosing for 4 hours on Days 1, 8, and 15 of each 28-day cycle

SUMMARY:
The purpose of the study was to assess efficacy, tolerability, safety and pharmacokinetics of Romidepsin in subjects with progressive or relapsed peripheral T-cell lymphoma

DETAILED DESCRIPTION:
This is a Phase 1/2, non-randomized, open-label, single-arm trial with two phases. The first phase is a 3 + 3 dose escalation phase to determine a recommended dose for treating patients with Peripheral T-Cell Lymphoma (PTCL) or Cutaneous T-Cell Lymphoma (CTCL) based on the assessment of Dose Limiting Toxicities (DLTs).The second phase will assess efficacy at the recommended dose by measuring objective response [Complete Response (CR), Unconfirmed Complete Response (CR(u)) or Partial Response (PR)] and determining best overall response of each patient. Phase 1 will enroll a maximum of 12 patients and Phase 2 will enroll up to approximately 40 patients

ELIGIBILITY:
Inclusion Criteria:

Patients must fulfill all of the following criteria to be eligible for study participation and have:

* Histologically confirmed Peripheral T cell Lymphoma (PTCL) Not Otherwise Specified (NOS), Angioimmunoblastic T-cell Lymphoma, enteropathy- type T-cell lymphoma, subcutaneous panniculitis-like T-cell lymphoma, cutaneous T-cell lymphoma (excludes mycosis fungoides or Sezary syndrome) , hepatosplenic T-cell lymphoma, Anaplastic Large cell lymphoma (ALCL) [anaplastic lymphoma kinase-1 (ALK-1) negative], patients with ALK 1 expressing ALCL (ALK-1 positive) who have relapsed disease after Autologous Stem-Cell Transplantation, Transformed mycosis fungoides (MF), or Sézary syndrome (SS);

  * Age ≥20 years;
  * Written informed consent;
  * Progressive Disease following at least one systemic therapy or refractory to at least one prior systemic therapy;
  * Eastern Cooperative Oncology Group (ECOG) performance status of 0-2;
  * Sufficient functions of bone marrow or other organs as evidenced by
* Hemoglobin ≥8.0 g/dL (The value after the 7th day of transfusion)
* Absolute neutrophil count (ANC) ≥1.0×10^9/L (The value after the 7th day of G-CSF)
* Platelet counts ≥100 x 10^9/L, or, if bone marrow infiltration is recognized, ≥75 ×10^9/L
* Total bilirubin (Total-Bil) ≤2 x upper limit of normal (ULN) (≤3.0 x ULN in the presence of demonstrable liver metastasis)
* Aspartate Aminotransferase (AST)/Serum Glutamic-Oxaloacetic Transaminase (SGOT) ≤2 x Upper Limit Normal (ULN) (≤3.0 x ULN in the presence of demonstrable liver metastasis)
* Alanine Aminotransferase (ALT)/Serum Glutamic-Oxaloacetic Transaminase (SGOT) ≤2 x ULN (≤3.0 x ULN in the presence of demonstrable liver metastasis)
* Serum creatinine ≤ 2 x ULN

  * Serum potassium ≥ lower limit of normal (LLN) and magnesium
  * Patients for whom at least 1 measurable lesion is confirmed in the lesion assessment before enrollment; and
  * Negative urine or serum pregnancy test on females of childbearing potential.

Exclusion Criteria: Confirmation should be made before enrollment, and the subjects corresponding to the criteria should not be enrolled.

1. Subjects in whom central nervous lymphoma is recognized during the screening period (If brain metastasis is suspected clinically, CT should be performed.)
2. Subjects undergoing chemotherapy or immunotherapy for the purpose of treatment of the target disease within 22 days before C1D1 (including C1D1) (using antibody drugs only within 3 months before C1D1)
3. Subjects receiving local application of steroids within 15 days before C1D1 (including C1D1) Use of steroids for the purpose other than that of treatment of the target disease should be allowed (Only CTCL subjects)
4. Subjects receiving systemic application of steroids within 22 days before C1D1 (including C1D1) (It is acceptable to continue the use of the steroid for the purpose of treatment of the target disease,which administered in doses ≤ 10mg/day prednisolone or equivalent dose of other glucocorticoid. However increase of steroid dose cannot be allowed during the study period)
5. Subjects undergoing radiation therapy, PUVA therapy or TSEB for the purpose of treatment of the target disease within 22 days before C1D1 (including C1D1)
6. Subjects using other investigational products within 22 days before C1D1 (including C1D1) (using antibody drugs only within 3 months before C1D1)
7. Subjects undergoing blood transfusion and using G-CSF within 8 days before C1D1 (including C1D1)
8. Subjects with the following abnormalities in the cardiac function

   1. Congenital QT prolongation syndrome
   2. QTc interval >480 msec
   3. Myocardial infarction within 6 months before C1D1. Subjects with a history of myocardial infarction between 6 and 12 months prior to C1D1 who are asymptomatic and have had a negative cardiac risk assessment (treadmill stress test, nuclear medicine stress test, or stress echocardiogram) since the event may occur
   4. Significant ECG abnormalities including atrio-ventricular (AV) block type II, 3rd degree AV block, or bradycardia (ventricular rate less than 50 beats/min)
   5. Symptomatic coronary artery disease (CAD) (e.g., Angina Canadian Class II-IV).
   6. An ECG recorded at screening showing significant ST depression (ST depression of ≥2 mm, measured from isoelectric line to the ST segment at a point 60 msec at the end of the QRS complex). If there is any doubt, the subject should have a stress imaging study and, if abnormal, angiography to define whether or not CAD is present.
   7. Congestive heart failure (CHF) that meets New York Heart Association (NYHA) Class II to IV definitions and/or ejection fraction <40% by MUGA scan or <50% by echocardiogram and/or MRI
   8. A known history of sustained ventricular tachycardia (VT), ventricular fibrillation (VF), torsade de pointes, or cardiac arrest unless currently addressed with an automatic implantable cardioverter defibrillator (AICD)
   9. Hypertrophic cardiomyopathy or restrictive cardiomyopathy from prior treatment or other causes (if there is any doubt, see ejection fraction criteria above)
   10. Uncontrolled hypertension, i.e., systolic blood pressure (BP) is greater than or equal to 160 mmHg or diastolic BP is greater than or equal to 95 mmHg; subjects who have a history of hypertension controlled by medication must be on a stable dose (for at least one month)
   11. Subjects with cardiac arrhythmia requiring an anti-arrhythmic drug
9. Concomitant use of a drug which may induce significant QT prolongation (refer to 9.2. Prohibited Concomitant Medications and Procedures.)
10. Concomitant use of strong or moderate CYP3A4 inhibitors which include grapefruit juice
11. Concomitant use of CYP3A4 inducers which include St John's Wort (1st step only)
12. Concomitant use of therapeutic warfarin which has a potential drug interaction. Use of a small dose of warfarin or other anticoagulant agent to maintain patency of venous access port and cannulas is permitted.
13. Clinically important active infections
14. Known infection with human immunodeficiency virus (HIV) antibody positive, HBs antigen positive or HCV antibody positive. If negative for HBsAg but HBcAb and/or HBsAb positive status, a HBV DNA test will be performed and if positive the subject will be excluded.
15. Subjects undergoing a wide range of radiation therapy in ≥30% of the bone marrow (such as all parts of the pelvic area or a half of the spinal cord) in the past. The subjects undergoing systemic radiation (including systemic electron therapy) as previous treatment for ASCT will be excluded.
16. Subjects undergoing a surgery within 15 days before C1D1 (including C1D1); however, even if more than 15 days have passed since the surgery, subjects without evidence of wound healing will be excluded.
17. Subjects who are during recovery process from severe wound or fracture.
18. Subjects with a history of allogeneic stem cell transplantation
19. Patients who are breast-feed during period of the IP administration or within 28 days after the end of the IP administration.
20. Subjects with a history of any other malignant tumor or solid cancer within previous 3 years (excluding basal or squamous cell carcinoma of skin, and in situ carcinoma of the cervix (CIN3) that has been treated curatively)
21. Subject with a history of hematological malignant tumor (other than T-cell lymphoma)
22. Subjects for whom transfusion of red blood cells or platelets is impossible (such as clinical state and religious beliefs)
23. Significant medical or psychiatric situation by which all of the study procedures may not be observed
24. Subjects receiving romidepsin in the past (Other HDAC inhibitors are acceptable)
25. Subjects judged to be inappropriate for this study by the investigator or sub-investigator.
26. Concomitant use of rifampicin.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 51 (Actual)
Dates: Start 2011-12-01 (Actual); Primary Completion 2015-07-28 (Actual); Study Completion 2018-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Toru Sasaki, Study Director — Celgene K.K.
Locations (17):
- Japan (17):
  - Nagoya Daini Red Cross Hospital, Nagoya, Aichi-ken
  - Nagoya City University Hospital, Nagoya, Aichi-ken
  - National Cancer Center Hospital East, Kashiwa, Chiba
  - Ehime University Hospital, Tōon, Ehime
  - Chugoku Central Hospital, Fukuyamashi, Hiroshima
  - Sapporo Hokuyu Hospital, Sapporo, Hokkaido
  - Sapporo Medical University Hospital, Sapporo, Hokkaido
  - Tokai University School of Medicine, Isehara, Kanagawa
  - Kochi Medical School Hospital, Nankoku, Kochi
  - Kinki University Hospital, Sayama, Osaka
  - National Cancer Center Hospital, Chūō, Tokyo
  - Japanese Red Cross Medical Center, Shibuya City, Tokyo
  - Kyushu University Hospital, Fukuoka
  - Kumamoto University Hospital, Kumamoto
  - University hospital, Kyoto prefectural University of Medicine, Kyoto
  - Tohoku University Hospital, Miyagi
  - The Cancer Institute Hospital of JFCR, Tokyo

REFERENCES:
- [Derived] Maruyama D, Tobinai K, Ogura M, Uchida T, Hatake K, Taniwaki M, Ando K, Tsukasaki K, Ishida T, Kobayashi N, Ishizawa K, Tatsumi Y, Kato K, Kiguchi T, Ikezoe T, Laille E, Ro T, Tamakoshi H, Sakurai S, Ohtsu T. Romidepsin in Japanese patients with relapsed or refractory peripheral T-cell lymphoma: a phase I/II and pharmacokinetics study. Int J Hematol. 2017 Nov;106(5):655-665. doi: 10.1007/s12185-017-2286-1. Epub 2017 Jun 29. PMID 28664499

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a Phase 1/2 open-label dose-escalation study. Phase 1 part composed of Cohort 1 (9mg/m^2) and Cohort 2 (14mg/m^2). Japanese participants were enrolled in order from Cohort 1. The dose used in the Phase 2 part was determined based on the frequency of dose limiting toxicities in Phase 1.
Pre-assignment Details: Those with relapsed, recurring or refractory peripheral T-cell lymphoma (PTCL) and cutaneous T-cell lymphoma (CTCL) were enrolled in the Phase 1 part of this study. In Phase 2, the target disease was relapsed, recurring or refractory PTCL only. Results are reported up to the data cut-off of 28 July 2015.
Groups:
- Phase 1: Romidepsin 9mg/m^2: Romidepsin 9mg/m^2 by intravenous (IV) infusion on Days 1, 8, 15 of each 28-day cycle
- Phase 1: Romidepsin 14mg/m^2; Phase 2: Romidepsin 14mg/m^2: Romidepsin 14mg/m^2 by intravenous (IV) infusion on Days 1, 8, 15 of each 28-day cycle.
Period: Phase 1 (First Step)
Arm/Group | Phase 1: Romidepsin 9mg/m^2 | Phase 1: Romidepsin 14mg/m^2 | Phase 2: Romidepsin 14mg/m^2
Started | 3 | 8 | 0
Completed | 1 (Completed = on treatment) | 1 (Completed = on treatment) | 0
Not Completed | 2 | 7 | 0
Not completed — Disease Progression | 1 | 1 | 0
Not completed — Withdrawal by Subject | 1 | 2 | 0
Not completed — Adverse Event | 0 | 3 | 0
Not completed — Other | 0 | 1 | 0
Period: Phase 2 (Second Step)
Arm/Group | Phase 1: Romidepsin 9mg/m^2 | Phase 1: Romidepsin 14mg/m^2 | Phase 2: Romidepsin 14mg/m^2
Started | 0 | 0 | 40
Completed | 0 | 0 | 7
Not Completed | 0 | 0 | 33
Not completed — Disease Progression | 0 | 0 | 17
Not completed — Adverse Event | 0 | 0 | 10
Not completed — Withdrawal by Subject | 0 | 0 | 4
Not completed — Protocol Violation | 0 | 0 | 1
Not completed — Other | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Intent to Treat (ITT) includes all participants who received at least one dose of romidepsin.
Groups:
- Total: Total of all reporting groups
Arm/Group | Phase 1: Romidepsin 9mg/m^2 | Phase 1: Romidepsin 14mg/m^2 | Phase 2: Romidepsin 14mg/m^2 | Total
Number analyzed (Participants) | 3 | 7 | 40 | 50
Age, Continuous [Mean (Standard Deviation); unit: years] | 59.0 (9.54) | 73.6 (4.20) | 68.5 (8.43) | 68.7 (8.47)
Age, Customized [Number; unit: participants]
  <65 years | 2 | 0 | 12 | 14
  ≥65 years | 1 | 7 | 28 | 36
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 17 | 21
  Male | 1 | 5 | 23 | 29
Disease Type by Investigator [Number; unit: participants] — PTCL is included in a heterogenous group of rare diseases resulting from clonal proliferation of mature thymic lymphocytes. These T-cell tumors account for about 10% to 15% of all lymphoid tumors. CTCL is a non-Hodgkin's lymphoma of helper T-cells that usually presents in the skin. It is classified mainly into mycosis fungoides and Sézary syndrome, and the stage is classified by the Tumor Node Metastasis Blood (TNMB) classification.
  participants
    PTCL | 2 | 6 | 40 | 48
    CTCL | 1 | 1 | 0 | 2
Eastern Cooperative Oncology Group (ECOG) [Number; unit: participants] — Eastern Cooperative Oncology Group (ECOG) performance status is used by doctors and researchers to assess how a participant's disease is progressing, assess how the disease affects the daily living activities of the participant and determine appropriate treatment and prognosis. 0 = Fully Active (Most Favorable Activity); 1 = Restricted activity but ambulatory; 2 = Ambulatory but unable to carry out work activities; 3 = Limited Self-Care; 4 = Completely Disabled, No self-care (Least Favorable Activity)
  participants
    0 = (Fully Active) | 0 | 4 | 22 | 26
    1 = (Restrictive but ambulatory) | 1 | 2 | 14 | 17
    2 = (Ambulatory but unable to work) | 2 | 1 | 4 | 7
    3 = (Limited self care) | 0 | 0 | 0 | 0
    4 = (Completely Disabled) | 0 | 0 | 0 | 0
Body Surface Area (BSA) [Mean (Standard Deviation); unit: m2] — BSA is the total surface area of the body and was used to calculate the dosage for romidepsin.
  m2 | 1.640 (0.1114) | 1.563 (0.2034) | 1.554 (0.1768) | 1.561 (0.1757)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Dose-limiting Toxicity (DLT) in Accordance With National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) Version 3.0 as Determined by the Efficacy and Safety Evaluation Committee (ESEC)
Description: DLT was defined as an adverse event (AE) occurring in Cycle 1 in Phase 1 and judged that the causal relationship to the investigational product could not be denied. The severity of all AEs was graded based upon the NCI CTCAE version 3.0. DLTs were defined as: • Grade 4 Hemoglobin <6.5 g/dL • Grade 4 Neutrophil <500/μL continuing for at least 5 days • Febrile neutropenia (Grade 4 neutropenia caused by fever and ≥ 38.5° C for more than 1 hour) • Grade 4 thrombocyte (< 25,000/μL), or thrombocytopenia with hemorrhage requiring platelet transfusion • Nausea, vomiting, or diarrhea at > grade 3 in spite of treatment • Grade 3 ALT (alanine aminotransferase) or AST (aspartate aminotransferase) values continued for 7 days. • Grade 4 ALT or AST • Grade 2 arrhythmia • Grade 4 non-hematological AEs • Other grade 3 non-hematological AEs except transient fatigue, anorexia, hyponatremia, and tumor lysis syndrome • Other AEs leading to discontinuation of administration
Time Frame: Up to Day 28; Cycle 1
Population: DLT population included all participants in the Phase 1 portion who received at least one dose of romidepsin. Of 8 participants enrolled in the 14mg/m^2 cohort, 2 participants, one with a critical Good Clinical Practice (GCP)violation and the other who did not complete Cycle 1 due to consent withdrawal, were excluded from the DLT assessment.
Measure: Number; unit: participants
Groups:
- Phase 1: Cohort 1: Romidepsin 9mg/m^2: Romidepsin 9mg/m^2 by intravenous (IV) infusion on Days 1, 8, 15 of each 28-day cycle
- Phase 1: Cohort 2: Romidepsin 14mg/m^2: Romidepsin 14mg/m^2 by intravenous (IV) infusion on Days 1, 8, 15 of each 28-day cycle.
Arm/Group | Phase 1: Cohort 1: Romidepsin 9mg/m^2 | Phase 1: Cohort 2: Romidepsin 14mg/m^2
Number analyzed (Participants) | 3 | 6
participants | 0 | 0

2. Primary Outcome: Percentage of PTCL Participants With an Overall Best Response in Accordance With a Modified International Workshop Response Criteria (IWC) 1999 in Phase 2
Description: Objective disease response in PTCL was defined as patients with a complete response (CR), unconfirmed complete response (CRu) or a partial response (PR) according to modified IWC 1999 criteria and assessed by an independent efficacy reviewer. A CR is >75% decrease in size of maximum 6 largest target within nodal and extranodal lesions, complete disappearance of other nodal and extranodal; total disappearance of clinical disease; disease-related signs and symptoms, normalization of biochemical abnormalities, disappearance of spleen, liver, or kidney enlargement; no bone marrow (BM) involvement, no new sites of disease. CRu: all above criteria fulfilled except for BM involvement is indeterminate. PR: a ≥50% decrease in size of 6 largest target lesions and no increase other nodal and extranodal; no progression of clinical disease; disease-related signs and symptoms, normalization or biochemical abnormalities, no progression in size of liver, spleen, or kidney; and no new sites of disease
Time Frame: Tumor assessments performed every 2 months; median follow-up time was 100 days; up to the data cut-off of 28 July 2015
Population: Intent to treat population for participants with PTCL who received at least one dose of Romidepsin
Measure: Number (95% Confidence Interval); unit: percentage of participants
Groups:
- Total: Romidepsin 14mg/m^2: Romidepsin 14mg/m^2 by intravenous (IV) infusion on Days 1, 8, 15 of each 28-day cycle.
Arm/Group | Phase 1: Romidepsin 9mg/m^2 | Phase 1: Romidepsin 14mg/m^2 | Phase 2: Romidepsin 14mg/m^2 | Total: Romidepsin 14mg/m^2
Number analyzed (Participants) | 2 | 6 | 40 | 46
percentage of participants | 0 [0.000 to 0.000] | 66.7 [28.947 to 100.000] | 42.5 [27.180 to 57.820] | 45.7 [31.258 to 60.046]
Statistical Analysis 1: Comparison: Phase 2: Romidepsin 14mg/m^2; Test type: Superiority or Other; p < 0.0001, Binomial test for dichotomized response — Based on one sample binomial test for dichotomized response proportion against the null hypothesis ( H0 p≤0.1)

3. Secondary Outcome: Participants With Treatment-Emergent Adverse Events (TEAEs) Associated With Romidepsin
Description: An adverse event (AE) is any noxious, unintended, or untoward medical occurrence that may appear or worsen during the course of a study. An AE that resulted in any of the outcomes was defined as a serious (SAE): • Death • Life-threatening event • An inpatient hospitalization or prolongation of existing hospitalization • Persistent or significant disability or incapacity; • Congenital anomaly or birth defect • Other important medical event The investigator judged the relationship of an AE to study drug based on the timing of the AE relative to drug administration and whether or not other drugs, therapeutic interventions, or underlying conditions could provide an explanation for the event. The severity of an AE was evaluated by the investigator according to Common Terminology Criteria for Adverse Events (CTCAE Version 3.0), Japanese Clinical Oncology Group (JCOG) where Grade 1 = Mild, Grade 2 = Moderate, Grade 3 = Severe, Grade 4 = Life-threatening and Grade 5 = Death.
Time Frame: Day 1 of study drug through 30 days after the last dose of study drug or discontinuation date; Up to data cut-off of 28 July 2015; maximum follow up time was 184.3 weeks
Population: Safety population includes all participants who received at least one dose of romidepsin
Measure: Number; unit: participants
Arm/Group | Phase 1: Romidepsin 9mg/m^2 | Phase 1: Romidepsin 14mg/m^2 | Phase 2: Romidepsin 14mg/m^2 | Total: Romidepsin 14mg/m^2
Number analyzed (Participants) | 3 | 7 | 40 | 47
participants
  Any 1 TEAE | 3 | 7 | 40 | 47
  TEAE related to any study drug | 3 | 7 | 40 | 47
  TEAE with CTCAE Grade 3 or greater | 3 | 6 | 37 | 43
  TEAE with CTCAE ≥Grade 3 related to study drug | 3 | 6 | 37 | 43
  ≥ 1 serious TEAE | 1 | 4 | 10 | 14
  Serious TEAE related to study drug | 0 | 4 | 6 | 10
  TEAE leading to discontinuation of study drug | 0 | 3 | 10 | 13
  TEAE related leading to discontinuation of drug | 0 | 3 | 9 | 12
  TEAE leading to dose held of study drug | 1 | 4 | 24 | 28
  Related TEAE leading to dose held of study drug | 1 | 3 | 22 | 25
  TEAE leading to dose reduction of study drug | 0 | 4 | 17 | 21
  Related TEAE leading to dose reduction of drug | 0 | 4 | 17 | 21
  TEAE leading to dose interruption of study drug | 1 | 4 | 23 | 27
  Related TEAE leading to dose interruption of drug | 1 | 3 | 22 | 25
  At least one TEAE with NCI CTCAE Grade 5 | 0 | 0 | 2 | 2

4. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to the Last Measurable Concentration (AUC0-t) of Romidepsin in Phase 1
Description: Area under the plasma concentration-time curve from time zero to the last quantifiable time point, calculated by the linear trapezoidal rule when concentrations are increasing and the logarithmic trapezoidal method when concentrations are decreasing.
Time Frame: Day 1 at Cycle 1; collected at 0 (pre-dose), 1, 2, 3, and 4 (at the end of administration) hours after the start of administration, 0.25 (15 minutes), 0.5 (30 minutes), 1, 2, 4, 6, 20, and 44 hours after the end of administration
Population: PK Population includes of all participants who had sufficient concentration-time data to enable the calculation of PK parameters for at least one PK day. For those who were determined to be noncompliant to receiving romidepsin, or for those with incomplete data, a decision to include the analysis was made on a case-by-case basis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 1: Cohort 1: Romidepsin 9mg/m^2 | Phase 1: Cohort 2: Romidepsin 14mg/m^2
Number analyzed (Participants) | 3 | 7
ng*h/mL | 1023.76 (66.7) | 2325.55 (35.3)

5. Secondary Outcome: Area Under the Plasma Concentration-time Curve From Time Zero to Infinity (AUC∞) of Romidepsin in Phase 1
Description: Area under the plasma concentration-time curve from time zero extrapolated to infinity (AUC∞) of romidepsin on Day 1; if possible the area under the concentration-time curve from time zero to infinity, calculated by the linear trapezoidal rule and extrapolated to infinity was calculated according to the following equation: AUC∞ = AUCt + (Ct/ λz ), where Ct is the last quantifiable concentration.
Time Frame: as for outcome 4
Population: PK Population consisted of all participants who had sufficient concentration-time data to enable the calculation of PK parameters for romidepsin for at least one PK day. For those who were determined to be noncompliant to receiving romidepsin, or for those with incomplete data, a decision to include the analysis was made on a case-by-case basis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 1: Cohort 1: Romidepsin 9mg/m^2 | Phase 1: Cohort 2: Romidepsin 14mg/m^2
Number analyzed (Participants) | 3 | 7
ng*h/mL | 1027.08 (66.6) | 2330.91 (35.2)

6. Secondary Outcome: Maximum Plasma Concentration (Cmax) of Romidepsin in Phase 1
Description: The maximum observed plasma concentration of romidepsin (Cmax) obtained directly from the observed concentration versus time data
Time Frame: as for outcome 4
Population: Pharmacokinetic (PK) Population includes of all participants who had sufficient concentration-time data to enable the calculation of PK parameters for at least one PK day. For those who were determined to be noncompliant to receiving romidepsin, or for those with incomplete data, a decision to include the analysis was made on a case-by-case basis.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1: Cohort 1: Romidepsin 9mg/m^2 | Phase 1: Cohort 2: Romidepsin 14mg/m^2
Number analyzed (Participants) | 3 | 7
ng/mL | 269.75 (48.9) | 593.47 (37.2)

7. Secondary Outcome: Time to Maximum Plasma Concentration of Romidepsin (Tmax) in Phase 1
Description: The time to first maximum observed plasma concentration of romidepsin after a single dose on Day 1.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1: Cohort 1: Romidepsin 9mg/m^2 | Phase 1: Cohort 2: Romidepsin 14mg/m^2
Number analyzed (Participants) | 3 | 7
hours | 4.02 [1.9 to 4.02] | 2.00 [1.00 to 4.1]

8. Secondary Outcome: Terminal Phase Half-life of Romidepsin (t½) in Phase 1
Description: The terminal phase half-life of romidepsin after a single dose on Day 1, calculated according to the following equation: t½ = 0.693/λz, where λz is the terminal phase rate constant.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Phase 1: Cohort 1: Romidepsin 9mg/m^2 | Phase 1: Cohort 2: Romidepsin 14mg/m^2
Number analyzed (Participants) | 3 | 7
hours | 9.52 (19.8) | 9.12 (11.6)

9. Secondary Outcome: Apparent Total Clearance of Romidepsin (CL/F) of Romidepsin in Phase 1
Description: The apparent total clearance of romidepsin after a single dose on Day 1, calculated as dose/AUC0-infinity.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: L/h
Arm/Group | Phase 1: Cohort 1: Romidepsin 9mg/m^2 | Phase 1: Cohort 2: Romidepsin 14mg/m^2
Number analyzed (Participants) | 3 | 7
L/h | 14.29 (60.8) | 9.31 (35.4)

10. Secondary Outcome: Apparent Volume of Distribution (Vz/F) of Romidepsin in Phase 1
Description: Apparent volume of distribution, was calculated according to the equation: Vd/F = (CL/F)/λz
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: Liters
Arm/Group | Phase 1: Cohort 1: Romidepsin 9mg/m^2 | Phase 1: Cohort 2: Romidepsin 14mg/m^2
Number analyzed (Participants) | 3 | 7
Liters | 196.24 (86.8) | 122.47 (40.4)

11. Secondary Outcome: AUC0-t, at Steady State (ss) of Romidepsin in Phase 1 at Cycle 1, Day 15
Description: Area under the plasma concentration-time curve from time zero to the last quantifiable time point at steady state, calculated by the linear trapezoidal rule when concentrations are increasing and the logarithmic trapezoidal method when concentrations are decreasing
Time Frame: Day 15 at Cycle 1; collected at 0 (pre-dose), 1, 2, 3, and 4 (at the end of administration) hours after the start of administration, 0.25 (15 minutes), 0.5 (30 minutes), 1, 2, 4, 6, 20, and 44 hours after the end of administration
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng*h/mL
Arm/Group | Phase 1: Cohort 1: Romidepsin 9mg/m^2 | Phase 1: Cohort 2: Romidepsin 14mg/m^2
Number analyzed (Participants) | 3 | 6
ng*h/mL | 1024.66 (78.1) | 1825.74 (25.8)

12. Secondary Outcome: Cmax, ss of Romidepsin in Phase 1 at Cycle 1, Day 15
Description: Maximum observed concentration in plasma at steady state
Time Frame: as for outcome 11
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ng/mL
Arm/Group | Phase 1: Cohort 1: Romidepsin 9mg/m^2 | Phase 1: Cohort 2: Romidepsin 14mg/m^2
Number analyzed (Participants) | 3 | 6
ng/mL | 250.05 (63.3) | 489.47 (31.2)

13. Secondary Outcome: Tmax,ss of Romidepsin in Phase 1 at Cycle 1, Day 15
Description: Observed time to first maximum plasma concentration at steady state
Time Frame: as for outcome 11
Population: as for outcome 4
Measure: Median (Full Range); unit: hours
Arm/Group | Phase 1: Cohort 1: Romidepsin 9mg/m^2 | Phase 1: Cohort 2: Romidepsin 14mg/m^2
Number analyzed (Participants) | 3 | 6
hours | 1.95 [1.9 to 3.9] | 2.94 [1.0 to 4.3]

14. Secondary Outcome: Terminal Phase Half-life of Romidepsin (t½) in Phase 1 at Cycle 1, Day 15
Description: The terminal phase half-life of romidepsin after a single dose on Day 15, calculated according to the following equation: t½ = 0.693/λz, where λz is the terminal phase rate constant.
Time Frame: as for outcome 11
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: hours
Arm/Group | Phase 1: Cohort 1: Romidepsin 9mg/m^2 | Phase 1: Cohort 2: Romidepsin 14mg/m^2
Number analyzed (Participants) | 3 | 6
hours | 8.77 (18.6) | 9.01 (15.8)

15. Secondary Outcome: AUC0-t, Accumulation Ratio of Romidepsin in Phase 1, Cycle 1
Description: Area under the plasma concentration-time curve from time zero to the last quantifiable time point; accumulation ratio calculated as AUC (0-t),ss/AUC (0-t)
Time Frame: Day 1 and Day 15 in Cycle 1; collected at 0 (pre-dose), 1, 2, 3, and 4 (at the end of administration) hours after the start of administration, 0.25 (15 minutes), 0.5 (30 minutes), 1, 2, 4, 6, 20, and 44 hours after the end of administration
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase 1: Cohort 1: Romidepsin 9mg/m^2 | Phase 1: Cohort 2: Romidepsin 14mg/m^2
Number analyzed (Participants) | 3 | 6
ratio | 1.00 (19.6) | 0.83 (24.3)

16. Secondary Outcome: Cmax Accumulation Ratio of Romidepsin in Phase 1, Cycle 1
Description: Cmax of Romidepsin: accumulation ratio based on Cmax calculated as Cmax,ss/Cmax
Time Frame: Day 1 and Day 15 in Cycle 1; collected at 0 (pre-dose), 1, 2, 3, and 4 (at end of administration) hours after the start of administration, 0.25, 0.5, 1, 2, 4, 6, 20, and 44 hours after the end of administration. Day 8, Cycle 1, samples collected at 0 hour
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: ratio
Arm/Group | Phase 1: Cohort 1: Romidepsin 9mg/m^2 | Phase 1: Cohort 2: Romidepsin 14mg/m^2
Number analyzed (Participants) | 3 | 6
ratio | 0.93 (15.3) | 0.86 (22.2)

17. Secondary Outcome: The Percentage of Participants With Abnormal Q-wave and T Wave Intervals
Description: The time from the start of the Q-wave to the end of the T-wave QTc intervals greater than 450 msec post-baseline performed by centralized reviewer. The Bazett's (QTcB) and Fridericia (QTcF) correction were used as the standard clinical correction for calculating the heart rate-corrected QTc interval
Time Frame: Median follow-up: 100 days; up to data cut-off of 28 July 2015
Population: The ECG population includes all participants who received romidepsin on Day 1 of Cycle 1 with at least one post-baseline QTc result
Measure: Number; unit: percentage of participants
Arm/Group | Phase 1: Romidepsin 9mg/m^2 | Phase 1: Romidepsin 14mg/m^2 | Phase 2: Romidepsin 14mg/m^2 | Total: Romidepsin 14mg/m^2
Number analyzed (Participants) | 3 | 7 | 40 | 47
percentage of participants
  QTcB >450 msec | 100 | 57.1 | 55.0 | 55.3
  QTcB >480 msec | 66.7 | 28.6 | 0.0 | 4.3
  QTcB >500 msec | 33.3 | 14.3 | 0.0 | 2.1
  QTcB increase from predose >30 msec | 66.7 | 57.1 | 10.0 | 17.0
  QTcB increase from predose >60 msec | 33.3 | 28.6 | 0.0 | 4.3
  QTcF >450 msec | 33.3 | 14.3 | 10.0 | 10.6
  QTcF >480 msec | 33.3 | 14.3 | 0.0 | 2.1
  QTcF >500 msec | 33.3 | 14.3 | 0.0 | 2.1
  QTcF increase from predose >30 msec | 66.7 | 57.1 | 10.0 | 17.0
  QTcF increase from predose >60 msec | 33.3 | 14.3 | 0.0 | 2.1

18. Secondary Outcome: Percentage of PTCL Participants With the Best Response in Accordance With the Modified 2007 International Workshop Response Criteria as Assessed by IER
Description: Objective disease response in PTCL was defined as achieving a CR or PR based on the Modified 2007 IWC. A CR = a complete disappearance of all disease; lymph node mass regression to normal size on computerized tomography (CT) scan or negative on positron emission tomography (PET); non-palpable splenic and disappearance of liver nodules; infiltrate cleared on repeat bone marrow (BM), immunohistochemistry negative. PR = a reduction of measurable lesions; ≥ 50% decrease in sum of the products of the greatest diameters (SPD) of up to 6 largest dominant masses, no enlargement in size of other nodes; ≥ 50% decrease in SPD and no increase in liver or spleen.
Time Frame: Tumor assessments performed every 2 months; median follow-up time was 100 days; up to the data cut-off of 28 July 2015
Population: Intent to treat population for participants with PTCL who received at least one dose of romidepsin
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Phase 1: Cohort 1: Romidepsin 9mg/m^2 | Phase 1: Cohort 2: Romidepsin 14mg/m^2 | Phase 2: Romidepsin 14mg/m^2 | Total: Romidepsin 14mg/m^2
Number analyzed (Participants) | 2 | 6 | 40 | 46
percentage of participants | 0 [0.000 to 0.000] | 16.7 [0.000 to 46.487] | 42.5 [27.180 to 57.820] | 39.1 [25.027 to 53.234]

19. Secondary Outcome: Time to Response (TTR) for PTCL Participants With at Least a PR Based on the Modified 1999 IWC as Assessed by IER
Description: TTR for PTCL was defined as the time in days from first dose date to the first date of objective disease response.
Time Frame: Median follow-up time was 100 days; up to the data cut-off of 28 July 2015
Population: Intent to treat population for participants with PTCL who received at least one dose of romidepsin and achieved a PR or better (CR, CRu or PR)
Measure: Median (Full Range); unit: days
Arm/Group | Phase 1: Romidepsin 14mg/m^2 | Phase 2: Romidepsin 14mg/m^2 | Total: Romidepsin 14mg/m^2
Number analyzed (Participants) | 4 | 17 | 21
days | 109.0 [51.0 to 812.0] | 56.0 [49.0 to 71.0] | 56.0 [49.0 to 812.0]

20. Secondary Outcome: Time to Response (TTR) for PTCL Participants With at Least a PR Based on the Modified 2007 IWC as Assessed by IER
Description: TTR for PTCL was defined as the time in days from first dose date to the first date of objective disease response.
Time Frame: Median follow-up time was 100 days; up to the data cut-off of 28 July 2015
Population: as for outcome 19
Measure: Median (Full Range); unit: days
Arm/Group | Phase 1: Romidepsin 14mg/m^2 | Phase 2: Romidepsin 14mg/m^2 | Total: Romidepsin 14mg/m^2
Number analyzed (Participants) | 1 | 17 | 18
days | 737.0 [737.0 to 737.0] | 56.0 [50.0 to 71.0] | 56.0 [50.0 to 737.0]

21. Secondary Outcome: Kaplan Meier Estimate of Duration of Response (DOR) for PTCL Responders Based on the Modified 1999 IWC as Assessed by the IER.
Description: DOR was defined as the number of days from the date of the first disease response (Complete, Unconfirmed Complete or Partial Response) until the date of progression, analyzed using Kaplan-Meier methods.
Time Frame: Median follow-up time was 100 days; up to the data cut-off of 28 July 2015
Population: as for outcome 19
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 1: Cohort 2: Romidepsin 14mg/m^2 | Phase 2: Romidepsin 14mg/m^2 | Total: Romidepsin 14mg/m^2
Number analyzed (Participants) | 4 | 17 | 21
days | 106.00 [62.00 to 843.00] | 337.00 [50.00 to NA] — Not estimable due to the low number of events | 337.00 [62.00 to 843.00]

22. Secondary Outcome: Kaplan Meier Estimate of Duration of Response (DOR) for PTCL Responders Based on the Modified 2007 IWC as Assessed by the IER.
Description: as for outcome 21
Time Frame: Median follow-up time was 100 days; up to the data cut-off of 28 July 2015
Population: as for outcome 19
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 1: Cohort 2: Romidepsin 14mg/m^2 | Phase 2: Romidepsin 14mg/m^2 | Total: Romidepsin 14mg/m^2
Number analyzed (Participants) | 1 | 17 | 18
days | 163.00 [NA to NA] — Not available = Not estimable due to the low number of events | 337.00 [60.00 to NA] — Not available = Not estimable due to the low number of events | 163.00 [60.00 to NA] — Not available = Not estimable due to the low number of events

23. Secondary Outcome: Kaplan Meier Estimate of Time to Progression (TTP) in PTCL Participants Based on the 1999 IWC as Assessed by IER
Description: Time to progression (≥50% increase from the nadir in the individual sum of the products of the diameters of any index lesion; the reappearance of pathology, enlargement of liver/spleen, or unequivocal progression of non-measurable disease or appearance of any new lesions) was defined as the duration from the date of the first study drug dose to the date of relapse or progression
Time Frame: Median follow-up time was 100 days; up to the data cut-off of 28 July 2015
Population: ITT includes all participants who received at least one dose of romidepsin
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 1: Cohort 1: Romidepsin 9mg/m^2 | Phase 1: Cohort 2: Romidepsin 14mg/m^2 | Phase 2: Romidepsin 14mg/m^2 | Total: Romidepsin 14mg/m^2
Number analyzed (Participants) | 2 | 6 | 40 | 46
days | 114.00 [NA to NA] — Not estimable due to the low number of events | 899.00 [112.00 to 899.00] | 170.00 [99.00 to 392.00] | 179.00 [101.00 to 392.00]

24. Secondary Outcome: Kaplan Meier (K-M) Estimate of Time to Progression (TTP) in PTCL Participants Based on the Modified 2007 IWC as Assessed by IER
Description: as for outcome 23
Time Frame: Median follow-up time was 100 days; up to the data cut-off of 28 July 2015
Population: ITT includes all participants who received at least one dose of romidepsin
Measure: Median (95% Confidence Interval); unit: days
Arm/Group | Phase 1: Cohort 1: Romidepsin 9mg/m^2 | Phase 1: Cohort 2: Romidepsin 14mg/m^2 | Phase 2: Romidepsin 14mg/m^2 | Total: Romidepsin 14mg/m^2
Number analyzed (Participants) | 2 | 6 | 40 | 46
days | NA [NA to NA] — Median time to progression based on K-M estimate had not been reached | 899.00 [NA to NA] — Not estimable due to low number of events | 179.00 [96.00 to 392.00] | 179.00 [96.00 to 392.00]

ADVERSE EVENTS:
Time Frame: Day 1 of study drug through 30 days after the last dose of study drug or discontinuation date; Up to data cut-off of 28 July 2015; maximum time exposed to study was 1290 days; maximum time on study treatment was 184.3 weeks
Arm/Group | Phase 1: Romidepsin 9mg/m^2 | Phase 1: Romidepsin 14mg/m^2 | Phase 2: Romidepsin 14mg/m^2 | Total: Romidepsin 14mg/m^2
Serious Adverse Events (participants affected / at risk) | 1/3 | 4/7 | 10/40 | 14/47
Other Adverse Events (participants affected / at risk) | 3/3 | 7/7 | 40/40 | 47/47
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Romidepsin 9mg/m^2 (N=3) | Phase 1: Romidepsin 14mg/m^2 (N=7) | Phase 2: Romidepsin 14mg/m^2 (N=40) | Total: Romidepsin 14mg/m^2 (N=47)
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 1 | 2
Bacterial infection (Infections and infestations) | 0 | 1 | 0 | 1
Hepatitis B (Infections and infestations) | 0 | 1 | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Pneumonia bacterial (Infections and infestations) | 0 | 0 | 1 | 1
Sepsis (Infections and infestations) | 0 | 0 | 1 | 1
Urinary tract infection (Infections and infestations) | 0 | 0 | 1 | 1
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 1
Cardiac failure acute (Cardiac disorders) | 0 | 0 | 1 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 1
Akathisia (Nervous system disorders) | 1 | 0 | 0 | 0
Altered state of consciousness (Nervous system disorders) | 0 | 1 | 0 | 1
Depressed level of consciousness (Nervous system disorders) | 0 | 0 | 1 | 1
Pyrexia (General disorders) | 0 | 0 | 2 | 2
Multi-organ failure (General disorders) | 0 | 0 | 1 | 1
Cancer pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Diffuse large B-cell lymphoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Retinal detachment (Eye disorders) | 0 | 0 | 1 | 1
Gastrointestinal haemorrhage (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 1 | 1
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 1 | 1
Hyperkalemia (Metabolism and nutrition disorders) | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Phase 1: Romidepsin 9mg/m^2 (N=3) | Phase 1: Romidepsin 14mg/m^2 (N=7) | Phase 2: Romidepsin 14mg/m^2 (N=40) | Total: Romidepsin 14mg/m^2 (N=47)
Thrombocytopenia (Blood and lymphatic system disorders) | 3 | 7 | 39 | 46
Lymphopenia (Blood and lymphatic system disorders) | 3 | 7 | 34 | 41
Leukopenia (Blood and lymphatic system disorders) | 3 | 6 | 33 | 39
Neutropenia (Blood and lymphatic system disorders) | 3 | 5 | 32 | 37
Anaemia (Blood and lymphatic system disorders) | 2 | 3 | 12 | 15
Nausea (Gastrointestinal disorders) | 3 | 4 | 20 | 24
Vomiting (Gastrointestinal disorders) | 3 | 3 | 15 | 18
Diarrhoea (Gastrointestinal disorders) | 2 | 2 | 14 | 16
Constipation (Gastrointestinal disorders) | 0 | 1 | 15 | 16
Stomatitis (Gastrointestinal disorders) | 0 | 2 | 6 | 8
Abdominal discomfort (Gastrointestinal disorders) | 0 | 1 | 1 | 2
Abdominal pain upper (Gastrointestinal disorders) | 1 | 0 | 1 | 1
Lip dry (Gastrointestinal disorders) | 2 | 0 | 0 | 0
Periodontal disease (Gastrointestinal disorders) | 0 | 0 | 2 | 2
Dental caries (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Gastritis (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Sensitivity of teeth (Gastrointestinal disorders) | 0 | 1 | 0 | 1
Pyrexia (General disorders) | 3 | 5 | 23 | 28
Fatigue (General disorders) | 3 | 1 | 12 | 13
Malaise (General disorders) | 0 | 3 | 10 | 13
Injection site reaction (General disorders) | 0 | 2 | 4 | 6
Oedema peripheral (General disorders) | 1 | 0 | 3 | 3
Chills (General disorders) | 0 | 0 | 2 | 2
Face oedema (General disorders) | 0 | 0 | 2 | 2
Hypothermia (General disorders) | 1 | 0 | 0 | 0
Influenza like illness (General disorders) | 1 | 0 | 0 | 0
Non-cardiac chest pain (General disorders) | 1 | 0 | 0 | 0
Decreased appetite (Metabolism and nutrition disorders) | 3 | 4 | 21 | 25
Hypokalaemia (Metabolism and nutrition disorders) | 1 | 2 | 7 | 9
Hypophosphataemia (Metabolism and nutrition disorders) | 0 | 1 | 9 | 10
Hyponatraemia (Metabolism and nutrition disorders) | 0 | 2 | 6 | 8
Hypermagnesaemia (Metabolism and nutrition disorders) | 1 | 1 | 4 | 5
Hypoalbuminaemia (Metabolism and nutrition disorders) | 0 | 1 | 5 | 6
Hypocalcaemia (Metabolism and nutrition disorders) | 1 | 1 | 4 | 5
Hyperkalaemia (Metabolism and nutrition disorders) | 0 | 1 | 4 | 5
Hypomagnesaemia (Metabolism and nutrition disorders) | 0 | 0 | 4 | 4
Dehydration (Metabolism and nutrition disorders) | 0 | 0 | 3 | 3
Hyperuricaemia (Metabolism and nutrition disorders) | 1 | 0 | 2 | 2
Tumour lysis syndrome (Metabolism and nutrition disorders) | 0 | 0 | 3 | 3
Hypercalcaemia (Metabolism and nutrition disorders) | 0 | 0 | 2 | 2
Haemoglobin decreased (Investigations) | 2 | 2 | 9 | 11
Alanine aminotransferase increased (Investigations) | 1 | 2 | 7 | 9
Weight decreased (Investigations) | 2 | 2 | 6 | 8
Aspartate aminotransferase increased (Investigations) | 0 | 1 | 8 | 9
Blood alkaline phosphatase increased (Investigations) | 1 | 0 | 3 | 3
Blood lactate dehydrogenase increased (Investigations) | 0 | 0 | 4 | 4
Electrocardiogram QT prolonged (Investigations) | 0 | 2 | 1 | 3
Blood phosphorus increased (Investigations) | 2 | 0 | 0 | 0
Blood urea increased (Investigations) | 1 | 0 | 1 | 1
Blood bilirubin increased (Investigations) | 0 | 1 | 0 | 1
Electrocardiogram ST-T change (Investigations) | 0 | 1 | 0 | 1
Electrocardiogram ST-T segment elevation (Investigations) | 0 | 1 | 0 | 1
Electrocardiogram T wave inversion (Investigations) | 0 | 1 | 0 | 1
Renal Function Test abnormal (Investigations) | 0 | 1 | 0 | 1
Dysgeusia (Nervous system disorders) | 3 | 4 | 24 | 28
Headache (Nervous system disorders) | 1 | 0 | 6 | 6
Peripheral Sensory neuropathy (Nervous system disorders) | 3 | 0 | 2 | 2
Akathisia (Nervous system disorders) | 1 | 0 | 0 | 0
Carotid arteriosclerosis (Nervous system disorders) | 0 | 1 | 0 | 1
Somnolence (Nervous system disorders) | 1 | 0 | 0 | 0
Rash (Skin and subcutaneous tissue disorders) | 0 | 1 | 4 | 5
Dry Skin (Skin and subcutaneous tissue disorders) | 0 | 0 | 2 | 2
Hyperhidrosis (Skin and subcutaneous tissue disorders) | 1 | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Haemorrhage subcutaneous (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Henoch-Schonlein purpura (Skin and subcutaneous tissue disorders) | 0 | 1 | 0 | 1
Rash macular (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1 | 3 | 2 | 5
Upper respiratory tract inflammation (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 4 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1 | 2
Hiccups (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pneumonitis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 1 | 1 | 3 | 4
Back Pain (Musculoskeletal and connective tissue disorders) | 1 | 2 | 2 | 4
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 1 | 0 | 2 | 2
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1
Periarthritis (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0 | 0
Nasopharyngitis (Infections and infestations) | 1 | 1 | 2 | 3
Influenza (Infections and infestations) | 1 | 1 | 1 | 2
Cytomegalovirus infection (Infections and infestations) | 0 | 1 | 1 | 2
Upper respiratory tract infection (Infections and infestations) | 1 | 0 | 1 | 1
Urinary Tract Infection (Infections and infestations) | 0 | 1 | 1 | 2
Bacterial Infection (Infections and infestations) | 0 | 1 | 0 | 1
Infected epidermal cyst (Infections and infestations) | 0 | 1 | 0 | 1
Infection (Infections and infestations) | 0 | 1 | 0 | 1
Pneumocystis jiroveci pneumonia (Infections and infestations) | 0 | 1 | 0 | 1
Atrial fibrillation (Cardiac disorders) | 0 | 1 | 3 | 4
Supraventriclar extrasystoles (Cardiac disorders) | 0 | 1 | 1 | 2
Angina pectoris (Cardiac disorders) | 0 | 1 | 0 | 1
Long QT syndrome (Cardiac disorders) | 1 | 0 | 0 | 0
Pericardial effusion (Cardiac disorders) | 0 | 1 | 0 | 1
Contusion (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Excoriation (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Fall (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Procedural Pain (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Phlebitis (Vascular disorders) | 1 | 2 | 1 | 3
Hypotension (Vascular disorders) | 2 | 1 | 0 | 1
Iritis (Eye disorders) | 0 | 1 | 0 | 1
Vitreous Floaters (Eye disorders) | 1 | 0 | 0 | 0
Proteinuria (Renal and urinary disorders) | 0 | 1 | 1 | 2
Pollakiuria (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hepatic function abnormal (Hepatobiliary disorders) | 0 | 0 | 3 | 3
Biliary colic (Hepatobiliary disorders) | 1 | 0 | 0 | 0
Hyperbilirubinaemia (Hepatobiliary disorders) | 0 | 1 | 0 | 1
Cancer Pain (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 2 | 2
Tumour associated fever (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 1
Insomnia (Psychiatric disorders) | 2 | 0 | 3 | 3
Gamma-glutamyltransferase increased (Investigations) | 0 | 1 | 0 | 1
Muscle Spasms (Musculoskeletal and connective tissue disorders) | 0 | 0 | 2 | 2
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Disclosure agreements vary; the Investigators shall not disclose any material/information disclosed by the Sponsor (Celgene KK) with the clinical trial or information obtained by conducting the clinical trial to third parties without Sponsor's prior written approval.